CLINICAL TRIAL: NCT01723904
Title: An Open-Label Study to Investigate the Safety and Efficacy of Rotigotine Add-On Therapy With Low Doses of Pramipexole or Ropinirole in Patients With Advanced Parkinson's Disease Phase 3B
Brief Title: A Phase 3b, Open-Label, Safety and Efficacy Study of Rotigotine as Add-On Therapy With Low Doses of Pramipexole or Ropinirole in Patients With Advanced Parkinson's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB BIOSCIENCES GmbH (Industry)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PD0015
Record Dates: First submitted 2012-11-06; First posted 2012-11-08 (Estimated); Results first posted 2014-06-03 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-05

CONDITIONS: Advanced Parkinson's Disease
Keywords: Rotigotine; Neupro
MeSH Terms: interventions — rotigotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rotigotine (Experimental): - Titration Period: Weekly titration to the subject's optimal dose of Rotigotine between 2 mg/24 h and 8 mg/24 h. In case of intolerable Adverse Events (AEs) one back-titration is allowed during the Titration Period.
  Duration of the Titration Period: Between 1 week and 5 weeks.
  - Maintenance Period: Starts once subject reached either optimal or maximal dose of Rotigotine. Subjects receive stable dose of Rotigotine throughout the Maintenance Period. No back-titration is allowed during the Maintenance Period.
  Duration of the Maintenance Period: Between 3 weeks and 7 weeks.
  Interventions: Drug: Rotigotine

INTERVENTIONS:
Drug: Rotigotine — Application of Rotigotine up to 8 mg/24 h patches for 24 hours.
  Other Names: Neupro

SUMMARY:
This study is to investigate the safety and efficacy of Rotigotine add-on therapy with low doses of Pramipexole or Ropinirole in patients with advanced-stage Parkinson's Disease (PD) who have insufficient response to L-dopa and low doses dopamine receptor agonists.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female, aged ≥ 30 and < 80 years at informed consent
* Subject has idiopathic Parkinson's Disease, of more than 3 years duration, as defined by the cardinal sign, bradykinesia, and the presence of at least 1 of the following: resting tremor, rigidity, impairment of postural reflexes, and without any known or suspected cause of Parkinsonism
* Subject has motor fluctuations such as wearing, dyskinesia
* Subject has experienced nocturias for at least 3 nights within 7 days prior to Baseline
* Subject is taking levodopa (L-DOPA, immediate and/or controlled release) in combination with benserazide or carbidopa and has been on a stable dose of L-DOPA for at least 28 days prior to Baseline (Visit 2)
* Subject is taking a non-ergot dopamine agonist (pramipexole ≤ 1.5 mg/day or ropinirole ≤ 6.0 mg/day) and has been on a stable dose of non-ergot dopamine agonist for at least 28 days prior to Baseline (Visit 2)

Exclusion Criteria:

* Subject is receiving therapy with tolcapone or budipine
* Subject is receiving therapy with one of the following drugs either concurrently or within 28 days prior to Baseline (Visit 2): alpha-methyl dopa, metoclopramide, reserpine, neuroleptics (except specific atypical neuroleptics: olanzapine, ziprasidone, aripiprazole, clozapine, quetiapine), monoamine oxidase A (MAO-A) inhibitors, methylphenidate, or amphetamine
* Subject has a history of symptomatic (not asymptomatic) orthostatic hypotension within the 6 months prior to Baseline (Visit 2)
* Subject has a known hypersensitivity to any components of the study medication, such as a history of significant skin hypersensitivity to adhesives, known hypersensitivity to other transdermal medications, or has unresolved contact dermatitis
* Subject is pregnant or nursing, or is of child-bearing potential (ie, is (i) not surgically sterile, or, (ii) not using adequate birth control methods [including at least one barrier method] or, (iii) not sexually abstinent, or (iv) not at least 2 years post menopausal)
* Subject had a previous diagnosis of narcolepsy, sleep apnea syndrome, restless legs syndrome, or periodic limb movement disorder

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-10; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (22):
- Australia (3):
  - 402, Chatswood, New South Wales
  - 401, Sydney, New South Wales
  - 403, Melbourne, Victoria
- Malaysia (3):
  - 202, Kuala Terengganu
  - 204, Kuching Sarawak
  - 201, Pulau Pinang
- Singapore (2):
  - 501, Singapore
  - 502, Singapore
- South Korea (11):
  - 104, Busan
  - 112, Busan
  - 109, Daegu
  - 111, Gyeonggi-do
  - 101, Seoul
  - 102, Seoul
  - 103, Seoul
  - 105, Seoul
  - 107, Seoul
  - 108, Seoul
  - 110, Seoul
- Taiwan (3):
  - 302, Taichung
  - 303, Tainan
  - 306, Taipei

REFERENCES:
- [Derived] Kim JM, Chung SJ, Kim JW, Jeon BS, Singh P, Thierfelder S, Ikeda J, Bauer L; Asia Pacific Rotigotine Add-on Study Group. Rotigotine transdermal system as add-on to oral dopamine agonist in advanced Parkinson's disease: an open-label study. BMC Neurol. 2015 Feb 28;15:17. doi: 10.1186/s12883-015-0267-7. PMID 25879416
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter study started to enroll subjects in 5 countries in October 2012.
Pre-assignment Details: Participant Flow refers to the Safety Set (SS). SS consists of all subjects who were enrolled and had at least 1 patch applied during the Treatment Period.
Groups:
- Rotigotine: - Titration Period: Weekly titration to the subject's optimal dose of Rotigotine between 2 mg/24 h and 8 mg/24 h. In case of intolerable Adverse Events (AEs) one back-titration is allowed during the Titration Period.
  Duration of the Titration Period: Between 1 week and 5 weeks.
  - Maintenance Period: Starts once subject reached either optimal or maximal dose of Rotigotine. Subjects receive stable dose of Rotigotine throughout the Maintenance Period. No back-titration is allowed during the Maintenance Period.
  Duration of the Maintenance Period: Between 3 weeks and 7 weeks.
  Rotigotine: Application of Rotigotine up to 8 mg/24 h patches for 24 hours.
Period: Overall Study
Arm/Group | Rotigotine
Started | 90
Completed | 79
Not Completed | 11
Not completed — Noncompliant | 3
Not completed — Adverse Event | 5
Not completed — Unable to follow protocol/ judged by inv | 3

BASELINE CHARACTERISTICS:
Population: Baseline characteristics refer to the Safety Set. The Safety Set consists of all subjects who had at least one patch application.
Arm/Group | Rotigotine
Number analyzed (Participants) | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (9.3)
Age, Customized [Number; unit: participants]
  < 65 years | 57
  >= 65 years | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 47
Region of Enrollment [Number; unit: participants]
  Taiwan | 8
  Malaysia | 6
  Singapore | 4
  Australia | 6
  Korea, Republic of | 66

OUTCOME MEASURES:

1. Primary Outcome: Clinical Global Impression (CGI) Item 4 (Side Effects) at the End of the Treatment Period
Description: The CGI Item 4 was used to assess side effects. It ranges from 0 to 4 as follows: 0 = Side effects not assessable
  1. = No side effects
  2. = Side effects do not significantly interfere with subject's functioning
  3. = Side effects significantly interfere with the subject's functioning
  4. = Side effects outweigh therapeutic efficacy.
Time Frame: Week 8 (Visit 8) of the 8 weeks Treatment Period (Titration and Maintenance Period)
Population: From the 90 subjects in the Safatey Set, 89 are included in the analysis of this outcome measure. Last Observation Carried Forward (LOCF) was used as a method of imputation for missing observations.
Measure: Number; unit: participants
Arm/Group | Rotigotine
Number analyzed (Participants) | 89
participants
  CGI Item 4 score of 1 | 61
  CGI Item 4 score of 2 | 22
  CGI Item 4 score of 3 | 3
  CGI Item 4 score of 4 | 3
  CGI Item 4 score of 3 or 4 | 6

2. Primary Outcome: Change From Baseline to the End of the Treatment Period in the Unified Parkinson's Disease Rating Scale (UPDRS) Part III ("on" State) Total Score
Description: The Unified Parkinson´s Disease Rating Scale Part III is an accepted and validated scale for the assessment of motor function in Parkinson´s disease. Each of the 27 sub-items in the UPDRS III is measured on a scale of 0 to 4, where 0 is normal and 4 represents severe abnormalities. The total scores therefore ranges from 0 to 108.
  A negative value in Change from Baseline to Week 8 indicates an improvement in motor functions from Baseline.
Time Frame: From Baseline (Week 0) to Week 8 (Visit 8) of the 8 weeks Treatment Period (Titration and Maintenance Period)
Population: Full Analysis Set (FAS) with Last Observation Carried Forward (LOCF) as a method of imputation for missing observations. FAS includes all subjects with at least 1 patch application during Treatment Period, and with an evaluable UPDRS Part III total score at Baseline and at least 1 valid value after Baseline to Day 64.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rotigotine
Number analyzed (Participants) | 89
units on a scale | -5.3 (8.3)

3. Primary Outcome: Change From Baseline to the End of the Treatment Period in the Unified Parkinson's Disease Rating Scale (UPDRS) Part II (Average of "on" and "Off" State) Total Score
Description: UPDRS Part II measures 'Activities in Daily Living'. The total score ranges from 0 (Best score possible) to 52 (Worst score possible).
  UPDRS Part II total score (average of "on" and "off" state) is the average of UPDRS Part II total score ("on" state) and Part II total score ("off" state).
  A negative value in Change from Baseline to Week 8 indicates an improvement in activities in daily living from Baseline.
Time Frame: From Baseline (Week 0) to Week 8 (Visit 8) of the 8 weeks Treatment Period (Titration and Maintenance Period)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rotigotine
Number analyzed (Participants) | 85
units on a scale | -1.5 (3.8)

4. Primary Outcome: Change From Baseline to the End of the Treatment Period in Absolute Time Spent "Off"
Description: Absolute time spent "off" is measured in hours per day. A negative value in Change from Baseline to Week 8 indicates that the time spent "off" decreased from Baseline and therefore indicates an improvement from Baseline.
  Only subjects with time spent "off" at Baseline (subset of the Full Analysis Set (FAS)) are included in the analysis of this outcome measure.
Time Frame: From Baseline (Week 0) to Week 8 (Visit 8) of the 8 weeks Treatment Period (Titration and Maintenance Period)
Population: Subjects with time spent "off" at Baseline in the FAS with Last Observation Carried Forward (LOCF) as a method of imputation for missing observations. FAS includes all subjects with at least 1 patch application during Treatment Period, and with an evaluable UPDRS Part III total score at Baseline and at least 1 valid value after Baseline to Day 64.
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | Rotigotine
Number analyzed (Participants) | 80
hours/day | -2.1 (2.9)

5. Secondary Outcome: Change From Baseline to the End of the Treatment Period in Time Spent "on" Without Troublesome Dyskinesia
Description: Absolute time spent "on" without troublesome dyskinesia is measured in hours per day. A positive value in Change from Baseline to Week 8 indicates that the time spent "on" without troublesome dyskinesia increased from Baseline and therefore indicates an improvement from Baseline.
Time Frame: From Baseline (Week 0) to Week 8 (Visit 8) of the 8 weeks Treatment Period (Titration and Maintenance Period)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | Rotigotine
Number analyzed (Participants) | 84
hours/day | 1.9 (3.1)

6. Secondary Outcome: Change From Baseline to the End of Treatment Period in Parkinson's Disease Sleep Scale 2 (PDSS-2) Total Score
Description: The Parkinson´s Disease Sleep Scale (PDSS) is a questionnaire with 15 questions to assess sleep disturbance and nocturnal disability in Parkinson´s disease. The item- scores can range between 0= never and 4= very often. The PDSS score is a sum score of all 15 questions.
  A negative value in Change from Baseline to Week 8 indicates an improvement from Baseline.
Time Frame: From Baseline (Week 0) to Week 8 (Visit 8) of the 8 weeks Treatment Period (Titration and Maintenance Period)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rotigotine
Number analyzed (Participants) | 89
units on a scale | -3.2 (7.5)

7. Secondary Outcome: Change From Baseline to the End of Treatment Period in the Pittsburgh Sleep Quality Index (PSQI) Global Score
Description: The Pittsburgh Sleep Quality Index (PSQI) is a questionnaire with 18 questions to assess sleep quality. The 18 questions are distributed to 7 elements with each element ranging from 0-3. The global score is the sum score of all 7 elements and ranges from 0-21 with higher values indicating worse sleep quality.
  A negative value in Change from Baseline to Week 8 indicates an improvement in sleep quality from Baseline.
Time Frame: From Baseline (Week 0) to Week 8 (Visit 8) of the 8 weeks Treatment Period (Titration and Maintenance Period)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rotigotine
Number analyzed (Participants) | 89
units on a scale | -0.7 (3.0)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected over the whole study duration from the Screening Period (Day -28 to Day -7) to the Safety Follow-up Visit (up to Day 78).
Description: Adverse Events refer to the Saftey Set. Safety Set consists of all subjects who were enrolled and had at least 1 patch applied during the Treatment Period.
Arm/Group | Rotigotine
Serious Adverse Events (participants affected / at risk) | 5/90
Other Adverse Events (participants affected / at risk) | 35/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotigotine (N=90)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotigotine (N=90)
Nausea (Gastrointestinal disorders) | 7 (9)
Application site pruritus (General disorders) | 12 (12)
Nasopharyngitis (Infections and infestations) | 5 (5)
Dizziness (Nervous system disorders) | 9 (11)
Dyskinesia (Nervous system disorders) | 7 (7)
Orthostatic hypotension (Vascular disorders) | 9 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days